CLINICAL TRIAL: NCT00305565
Title: Randomized Comparison of Outcomes in Patients With Treatment-Resistant Depression Who Receive VNS Therapy Administered at Different Amounts of Electrical Charge
Brief Title: Study Comparing Outcomes for Patients With Treatment Resistant Depression Who Receive VNS Therapy at Different Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-21-US
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: Depression; Chronic Depression; Bipolar Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Other)
  Interventions: Device: VNS Therapy
- Medium Dose (Other)
  Interventions: Device: VNS Therapy
- High Dose (Other)
  Interventions: Device: VNS Therapy

INTERVENTIONS:
Device: VNS Therapy — Received output current of 0.25 milliamps (mA)
  Other Names: VNS Therapy System
  Arms: Low Dose
Device: VNS Therapy — Received output current of 0.5-1.0 mA
  Other Names: VNS Therapy System
  Arms: Medium Dose
Device: VNS Therapy — Received output current of 1.0-1.5 mA
  Other Names: VNS Therapy System
  Arms: High Dose

SUMMARY:
This is a postmarket medical device study. The objective of this study is to compare the safety and effectiveness of Vagus Nerve Stimulation (VNS) Therapy administered at different amounts of electrical charge for the treatment of patients with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
This is a postmarket medical device study. This study will examine treatment outcomes for patients with TRD who are randomized to VNS Therapy administered at different amounts of electrical charge. The Sponsor, Cyberonics, provides funding for this study. Patients are followed for 54 weeks, 50 of those weeks are following implantation of the VNS Therapy system. No study sites will be permitted to enroll study subjects until Institutional Review Board (IRB) approval has been received. Sites are permitted to be approved by a local or a central IRB.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of chronic or recurrent depression and is currently experiencing a major depressive episode.
* Patient has not had an adequate response to four or more adequate antidepressant treatments from at least two different antidepressant treatment categories.
* Patient has (in the investigator's judgment) sufficient impairment from his/her depression and/or depression treatment that the potential benefits/risks of VNS Therapy are warranted.
* Patient must currently be receiving at least one antidepressant treatment; the patient must be receiving all current antidepressant treatments in a stable regimen.
* If the patient has a current diagnosis of bipolar disorder, the patient must be receiving a mood stabilizer.
* Patient must be 18 years of age or older and of legal age of consent.
* Patient must be able to complete the evaluations specified in the study procedures flow chart.
* Patient must provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.

Exclusion Criteria:

* Patient has had a bilateral or left cervical vagotomy.
* Patient currently uses, or is expected to use during the study, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
* A VNS Therapy System implant would pose an unacceptable surgical or medical risk for the patient.
* Patient is expected to require full body magnetic resonance imaging during the clinical study.
* Patient is acutely suicidal.
* Patient has a history of schizophrenia, schizoaffective disorder, or other psychotic disorder or a current major depressive episode that includes psychotic features (commonly referred to as psychotic depression).
* Patient has a history of rapid cycling bipolar disorder or a current diagnosis of bipolar disorder mixed phase.
* Patient has a history of borderline personality disorder.
* Patient has a history of drug or alcohol dependence within the 12 months prior to the baseline visit or currently takes a narcotic drug five or more days per week.
* Patient is currently enrolled in another investigational study.
* Patient has had a prior VNS Therapy System implant.

Note: Some IRBs may require additional conditions for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bunker, PharmD, Study Director — Cyberonics, Inc.
Locations (26):
- United States (26):
  - University of Arizona, Tucson, Arizona
  - Sutter Institute for Medical Research, Sacramento, California
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Evanston Northwestern Hospital, Evanston, Illinois
  - Clinical Research Institute, Wichita, Kansas
  - Brentwood Research Institute, Shreveport, Louisiana
  - Sheppard Pratt Hospital, Baltimore, Maryland
  - Pharmasite Research Inc., Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Psychiatric Recovery, Saint Paul, Minnesota
  - St. Louis University, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Community Clinical Research, Inc., Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Claghorn-Lesem Research Clinic, LTD, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Center for Anxiety and Depression, Mercer Island, Washington

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Murray CJ, Lopez AD. Evidence-based health policy--lessons from the Global Burden of Disease Study. Science. 1996 Nov 1;274(5288):740-3. doi: 10.1126/science.274.5288.740. No abstract available. PMID 8966556
- [Background] Geddes LA, Baker LE: Principles of Applied Biomedical Instrumentation, third edition. New York; John Wiley & Sons, 1989; 458-461.
- [Background] Rush AJ, Sackeim HA, Marangell LB, George MS, Brannan SK, Davis SM, Lavori P, Howland R, Kling MA, Rittberg B, Carpenter L, Ninan P, Moreno F, Schwartz T, Conway C, Burke M, Barry JJ. Effects of 12 months of vagus nerve stimulation in treatment-resistant depression: a naturalistic study. Biol Psychiatry. 2005 Sep 1;58(5):355-63. doi: 10.1016/j.biopsych.2005.05.024. PMID 16139581
- [Background] George MS, Rush AJ, Marangell LB, Sackeim HA, Brannan SK, Davis SM, Howland R, Kling MA, Moreno F, Rittberg B, Dunner D, Schwartz T, Carpenter L, Burke M, Ninan P, Goodnick P. A one-year comparison of vagus nerve stimulation with treatment as usual for treatment-resistant depression. Biol Psychiatry. 2005 Sep 1;58(5):364-73. doi: 10.1016/j.biopsych.2005.07.028. PMID 16139582
- [Background] Rush AJ, Marangell LB, Sackeim HA, George MS, Brannan SK, Davis SM, Howland R, Kling MA, Rittberg BR, Burke WJ, Rapaport MH, Zajecka J, Nierenberg AA, Husain MM, Ginsberg D, Cooke RG. Vagus nerve stimulation for treatment-resistant depression: a randomized, controlled acute phase trial. Biol Psychiatry. 2005 Sep 1;58(5):347-54. doi: 10.1016/j.biopsych.2005.05.025. PMID 16139580
- [Result] Aaronson ST, Carpenter LL, Conway CR, Reimherr FW, Lisanby SH, Schwartz TL, Moreno FA, Dunner DL, Lesem MD, Thompson PM, Husain M, Vine CJ, Banov MD, Bernstein LP, Lehman RB, Brannon GE, Keepers GA, O'Reardon JP, Rudolph RL, Bunker M. Vagus nerve stimulation therapy randomized to different amounts of electrical charge for treatment-resistant depression: acute and chronic effects. Brain Stimul. 2013 Jul;6(4):631-40. doi: 10.1016/j.brs.2012.09.013. Epub 2012 Oct 23. PMID 23122916

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 331 subjects at 29 sites were actually enrolled and implanted with the Vagus Nerve Stimulation (VNS) Therapy System, and were included in the safety dataset. Twenty-one subjects were excluded from the intent-to-treat (ITT) dataset, leaving 310 in the ITT population.
Groups:
- Low Dose: Received output current 0.25 milliamps (mA)
- Medium Dose: Received output current 0.5-1.0 mA
- High Dose: Received output current 1.0-1.5 mA
Period: Overall Study (Safety Population)
Arm/Group | Low Dose | Medium Dose | High Dose
Started | 111 | 107 | 113
Completed | 97 | 95 | 106
Not Completed | 14 | 12 | 7
Period: Overall Study (ITT Population)
Arm/Group | Low Dose | Medium Dose | High Dose
Started | 102 | 101 | 107
Completed | 89 | 90 | 102
Not Completed | 13 | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Low Dose: Received output current 0.25 mA
- Total: Total of all reporting groups
Arm/Group | Low Dose | Medium Dose | High Dose | Total
Number analyzed (Participants) | 102 | 101 | 107 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (10.5) | 47.2 (11.0) | 47.4 (10.8) | 47.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 69 | 73 | 210
  Male | 34 | 32 | 34 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 97 | 96 | 104 | 297
  Asian | 3 | 1 | 0 | 4
  African-American | 2 | 3 | 3 | 8
  Hispanic | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 102 | 101 | 107 | 310
Unipolar or Bipolar Depression [Number; unit: participants]
  Unipolar Depression (Single Episode) | 6 | 10 | 15 | 31
  Unipolar Depression (Recurrent) | 76 | 71 | 66 | 213
  Bipolar Depression | 20 | 20 | 26 | 66
Lifetime Episodes of Depression [Number; unit: participants] — This study specific characteristic data was not available for 1 participant in the Medium Dose Group.
  participants
    0-2 Episodes | 16 | 17 | 28 | 61
    3-5 Episodes | 23 | 21 | 22 | 66
    6-10 Episodes | 13 | 16 | 18 | 47
    >10 Episodes | 50 | 46 | 39 | 135
Duration of Illness [Mean (Standard Deviation); unit: Years] | 29.8 (12.1) | 26.3 (10.9) | 27.0 (12.1) | 27.7 (11.8)
Length of Current Major Depressive Episode [Mean (Standard Deviation); unit: Months] | 106.7 (122.8) | 106.1 (107.3) | 111.3 (146.3) | 108.1 (126.5)

OUTCOME MEASURES:

1. Primary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Mean Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
Time Frame: From Baseline to Study Week 22
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: repeated measures IDS-C observations
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 102 | 101 | 107
Number analyzed (repeated measures IDS-C observations) | 396 | 390 | 417
units on a scale | -9.96 (0.99) | -10.29 (1.00) | -10.30 (0.97)
Statistical Analysis 1: Comparison: Low Dose vs High Dose; The primary analysis consisted of contrasts comparing High Dose vs. Low Dose and Medium Dose vs. Low Dose averaged over the 4 Acute Phase visits using the Hochberg approach to adjust for multiplicity. If both comparisons involving the Low Dose were significant, then a test of High Dose vs. Medium Dose was evaluated at the P≤0.05 level. The pivotal analysis was performed on the ITT population using the last-observation-carried-forward (LOCF) approach to impute missing data; Test type: Superiority or Other; p = 0.803, Mixed Models Analysis; Mean Difference (Net) = 0.34, 95% CI 2-sided [-2.34 to 3.02]
Statistical Analysis 2: Comparison: Low Dose vs Medium Dose; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.813, Mixed Models Analysis; Mean Difference (Net) = 0.33, 95% CI 2-sided [-2.39 to 3.05]

2. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Percent Responders From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C percent of responders at week 22. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
percentage of participants | 16.5 | 17.5 | 21.0

3. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Percent Remitters From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C percent of remitters at week 22. Remission was defined as a score of less than or equal to 14 on the IDS-C.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
percentage of participants | 6.2 | 9.3 | 11.4

4. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Percent Responders From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C percent of responders at week 50. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 27.0 | 38.9 | 27.5

5. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Percent Sustained Responders at Study Week 50 (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  Sustained Response is defined as the percentage of Acute Phase responders (week 22) who were also responders at the end of the Long-term (week 50) phase. An analysis of sustained response was performed using the IDS-C to evaluate the long-term durability of the improvements in depression scores observed with adjunctive VNS Therapy.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 16 | 17 | 22
percentage of participants | 43.8 | 88.2 | 81.8

6. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Percent Remitters From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C percent of remitters at week 50. Remission was defined as a score of less than or equal to 14 on the IDS-C.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 14.6 | 15.6 | 17.6

7. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Percent Responders From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C percent of responders at week 22. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
percentage of participants | 20.6 | 21.6 | 23.8

8. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Percent Remitters From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C percent of remitters at week 22. Remission was defined as a score of less than or equal to 5 on the QIDS-C.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
percentage of participants | 6.2 | 9.3 | 9.5

9. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Percent Responders From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C percent of responders at week 50. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 36.0 | 44.4 | 34.3

10. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Percent Remitters From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C percent of remitters at week 50. Remission was defined as a score of less than or equal to 5 on the QIDS-C.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 15.7 | 16.7 | 16.7

11. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Percent Responders From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS percent of responders at week 22. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
percentage of participants | 16.5 | 25.8 | 28.6

12. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Percent Remitters From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS percent of remitters at week 22. Remission was defined as a score of less than or equal to 9 on the MADRS.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
percentage of participants | 5.2 | 11.3 | 11.4

13. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Percent Responders From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS percent of responders at week 50. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 36.0 | 47.8 | 37.3

14. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Percent Sustained Responders at Study Week 50 (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  Sustained Response is defined as the percentage of Acute Phase responders (week 22) who were also responders at the end of the Long-term (week 50) phase. An analysis of sustained response was performed using the MADRS to evaluate the long-term durability of the improvements in depression scores observed with adjunctive VNS Therapy.
Time Frame: From Baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 16 | 25 | 30
percentage of participants | 68.8 | 92.0 | 76.7

15. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Percent Remitters From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS percent of remitters at week 50. Remission was defined as a score of less than or equal to 9 on the MADRS.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 22.5 | 21.1 | 22.5

16. Secondary Outcome: Clinical Global Impressions Improvement Scale (CGI-I) Percent Response at Week 22 of the Acute Phase (ITT Population)
Description: Originally, the Clinical Global Impressions-Improvement (CGI-I) (Guy W 1976)was designed as a 7-item scale used to assess how much the patient's illness had improved or worsened relative to a baseline state at the beginning of the intervention.(1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
  In this study, the CGI-I was categorized into just two groups. A value of 1 (considered a response) was assigned for very much improved (at least 85% improvement) & much improved (at least 60% improvement). A value of 0 (considered non-response) was assigned for: minimally improved (at least 20-25% improvement), no change (between ±15% change), minimally worse (at least 20-55% worse), much worse (at least 60% worse), and very much worse (at least 80% worse). No score was assigned if the investigator did not provide a categorical rating at a particular follow-up visit.
Time Frame: At Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 96 | 105
percentage of participants | 20.6 | 28.1 | 31.4

17. Secondary Outcome: Clinical Global Impressions Improvement Scale (CGI-I) Percent Response at Week 50 of the Long-term Phase (ITT Population).
Description: as for outcome 16
Time Frame: At Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
percentage of participants | 41.6 | 53.3 | 48.0

18. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Percent Responders From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR percent of responders at week 22. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 95 | 96 | 105
percentage of participants | 9.5 | 15.6 | 19.0

19. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Percent Remitters From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR percent of remitters at week 22. Remission was defined as a score of less than or equal to 14 on the IDS-C.
Time Frame: From baseline to Study Week 22
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 95 | 96 | 105
percentage of participants | 5.3 | 9.4 | 11.4

20. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Percent Responders From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR percent of responders at week 50. Response was defined as greater than or equal to 50% improvement from baseline.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 88 | 88 | 101
percentage of participants | 28.4 | 36.4 | 26.7

21. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Percent Remitters From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR percent of remitters at week 50. Remission was defined as a score of less than or equal to 14 on the IDS-C.
Time Frame: From baseline to Study Week 50
Measure: Number; unit: percentage of participants
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 88 | 88 | 101
percentage of participants | 17.0 | 17.0 | 14.9

22. Post Hoc Outcome: Regression Analysis of Change in IDS-C Score vs. Total Charge Delivered Per Day
Description: Mixed models multivariate regression model was fitted for the outcome change from baseline IDS-C score as a function of log dose, where dose is measured by millicoulombs (mC), adjusting for other important covariates (e.g., visit number, total number of major depressive episodes, prior electroconvulsive therapy (ECT) history, total number of adequate drug trials and prior medication regimen).
  The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
Time Frame: 50 Weeks
Population: 50 Week Completers
Measure: Least Squares Mean (Standard Error); unit: Units on a scale per log(mC/Day)
Groups:
- Log Dose-Response Regression Coefficient: All dosing groups
Arm/Group | Log Dose-Response Regression Coefficient
Number analyzed (Participants) | 314
Units on a scale per log(mC/Day) | -4.91 (1.34)

23. Post Hoc Outcome: Regression Analysis of Change in MADRS Score vs. Total Charge Delivered Per Day
Description: Mixed models multivariate regression model was fitted for the outcome change from baseline MADRS score as a function of log dose, where dose is measured by millicoulombs (mC), adjusting for other important covariates (e.g., visit number, total number of major depressive episodes, prior ECT history, total number of adequate drug trials and prior medication regimen).
  The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
Time Frame: 50 Weeks
Population: 50 Week Completers
Measure: Least Squares Mean (Standard Error); unit: Units on a scale per log(mC/Day)
Arm/Group | Log Dose-Response Regression Coefficient
Number analyzed (Participants) | 314
Units on a scale per log(mC/Day) | -2.17 (0.93)

24. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Mean Percent Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C mean percent change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
mean percent change | -22.3 (25.3) | -24.9 (28.9) | -25.4 (31.4)

25. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Mean Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C mean change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
units on a scale | -16.9 (13.9) | -17.0 (14.6) | -15.3 (12.9)

26. Secondary Outcome: Inventory of Depressive Symptomatology-Clinician Administered (IDS-C) Mean Percent Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-C mean percent change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
mean percent change | -36.6 (28.8) | -36.5 (32.5) | -34.6 (30.7)

27. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Mean Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C mean change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
units on a scale | -4.4 (5.0) | -5.0 (5.4) | -4.7 (5.3)

28. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Mean Percent Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C mean percent change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
mean percent change | -23.7 (27.4) | -26.5 (29.8) | -26.3 (31.6)

29. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Mean Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C mean change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
units on a scale | -7.1 (5.7) | -7.2 (6.2) | -6.7 (5.1)

30. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Clinician Administered (QIDS-C) Mean Percent Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 16-item Inventory of Depressive Symptomatology (QIDS) (Rush et al. 2003) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 27. Higher values are considered to be worse outcomes.
  The QIDS-C mean percent change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
mean percent change | -37.9 (30.2) | 38.5 (32.8) | 38.2 (30.6)

31. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS mean change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
units on a scale | -8.4 (8.8) | -9.1 (10.7) | -9.6 (11.0)

32. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Percent Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS mean percent change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 97 | 97 | 105
mean percent change | -25.0 (26.1) | -26.7 (31.3) | 28.2 (33.5)

33. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS mean change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
units on a scale | -13.5 (11.6) | -14.3 (11.6) | -13.7 (10.8)

34. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Percent Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 10-item Montgomery-Asberg Scale (Montgomery and Asberg 1979) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 60. Higher values are considered to be worse outcomes.
  The MADRS mean percent change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 89 | 90 | 102
mean percent change | -39.3 (33.8) | -42.0 (34.2) | -40.8 (33.4)

35. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Mean Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR mean change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 95 | 96 | 105
units on a scale | -9.0 (11.4) | -11.1 (13.9) | -10.2 (13.7)

36. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Mean Percent Change From Baseline to Week 22 of the Acute Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR mean percent change at week 22
Time Frame: From baseline to Study Week 22
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 95 | 96 | 105
mean percent change | -19.6 (24.7) | -22.6 (29.4) | -22.7 (31.1)

37. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Mean Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR mean change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 88 | 88 | 101
units on a scale | -15.9 (15.0) | -16.7 (15.0) | -14.5 (13.5)

38. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDS-SR) Mean Percent Change From Baseline to Week 50 of the Long-term Phase (ITT Population).
Description: The 30-item Inventory of Depressive Symptomatology (IDS-C/SR) (Rush et al. 1986, 1996) is designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  The IDS-SR mean percent change at week 50
Time Frame: From baseline to Study Week 50
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 88 | 88 | 101
mean percent change | -33.5 (29.6) | -35.5 (32.2) | -32.4 (31.3)

ADVERSE EVENTS:
Time Frame: 54 Weeks
Arm/Group | Low Dose | Medium Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 31/111 | 19/107 | 16/113
Other Adverse Events (participants affected / at risk) | 103/111 | 104/107 | 111/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=111) | Medium Dose (N=107) | High Dose (N=113)
Body as a Whole (General disorders) | 19 | 9 | 13
Cardiovascular System (Cardiac disorders) | 1 | 1 | 1
Digestive System (Gastrointestinal disorders) | 3 | 1 | 1
Endocrine System (Endocrine disorders) | 0 | 1 | 0
Nervous System (Nervous system disorders) | 9 | 10 | 4
Respiratory System (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Skin and Appendages System (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urogenital System (Renal and urinary disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=111) | Medium Dose (N=107) | High Dose (N=113)
Body as a Whole (General disorders) | 80 | 78 | 92
Cardiovascular System (Cardiac disorders) | 12 | 13 | 15
Digestive System (Gastrointestinal disorders) | 37 | 45 | 47
Endocrine System (Endocrine disorders) | 4 | 0 | 1
Hemic System (Blood and lymphatic system disorders) | 4 | 2 | 2
Metabolic System (Metabolism and nutrition disorders) | 7 | 9 | 14
Musculoskeletal System (Musculoskeletal and connective tissue disorders) | 6 | 12 | 11
Nervous System (Nervous system disorders) | 73 | 62 | 85
Respiratory System (Respiratory, thoracic and mediastinal disorders) | 87 | 97 | 99
Skin and Appendages System (Skin and subcutaneous tissue disorders) | 9 | 7 | 6
Special Senses System (Ear and labyrinth disorders) | 11 | 6 | 15
Urogenital System (Renal and urinary disorders) | 8 | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less